CLINICAL TRIAL: NCT04819841
Title: A Phase I/II Study of Nula-cel in Autologous CD34+ Hematopoietic Stem Cells to Convert HbS to HbA for Treating Severe Sickle Cell Disease
Brief Title: Gene Correction in Autologous CD34+ Hematopoietic Stem Cells (HbS to HbA) to Treat Severe Sickle Cell Disease
Acronym: Restore
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kamau Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KMAU-001-001
Record Dates: First submitted 2021-03-24; First posted 2021-03-29 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Sickle Cell Disease
Keywords: sickle cell disease; sickle cell anemia; gene correction; gene therapy; CRISPR
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- nula-cel Drug Product (Experimental): nula-cel Drug Product is a human autologous CRISPR-Cas9 edited and sickle mutation-corrected HSPC product.
  Interventions: Genetic: nula-cel Drug Product

INTERVENTIONS:
Genetic: nula-cel Drug Product — nula-cel is administered via IV infusion following a myeloablative conditioning regimen

SUMMARY:
This study is a first-in-human, single-arm, open-label Phase I/II study of nula-cel in approximately 15 participants, diagnosed with severe Sickle Cell Disease. The primary objective is to evaluate safety of the treatment in this patient population, as well as preliminary efficacy and pharmacodynamic data.

DETAILED DESCRIPTION:
Participants diagnosed with severe SCD will receive nula-cel via IV infusion following myeloablative conditioning in an autologous HSCT setting.

ELIGIBILITY:
Inclusion Criteria:

* ≥12 to ≤ 40 years
* Severe disease, as defined by having experienced at least one of the following SCD-related events despite appropriate supportive care measures:
* recurrent severe VOC (≥ 4 episodes in the preceding 2 years)
* ACS (≥ 2 episodes in the prior 2 years with at least one episode in the past year)
* Lansky/Karnofsky performance status of ≥ 80

Exclusion Criteria:

* Available 10/10 HLA-matched sibling donor
* Prior HSCT or gene therapy
* Prior or current malignancy or myeloproliferative or a significant coagulation or immunodeficiency disorder
* Clinically significant and active bacterial, viral, fungal or parasitic infection
* Pregnancy or breastfeeding in a postpartum female
* Presence of a chromosomal abnormality/mutation that may put the participant at an increased risk for MDS or AML per investigator's judgment

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Estimated)
Dates: Start 2021-11-15 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who reach neutrophil engraftment | 42 days post-infusion
Incidence rate of treatment-related mortality | 100 days post-infusion
Incidence rate of treatment-related mortality | 12 months post-infusion
Overall survival | 24 months post-infusion
Frequency and severity of AEs/SAEs | 24 months post-infusion

SECONDARY OUTCOMES:
Time to neutrophil engraftment | through study completion, up to 24 months post-infusion
Time to platelet engraftment | through study completion, up to 24 months post-infusion
Evaluation of gene correction levels in peripheral myeloid cells | through study completion, up to 24 months post-infusion
Evaluation of adult Hgb as a percentage of total Hgb | through study completion, up to 24 months post-infusion
Evaluation of HbS as a percentage of total Hgb | through study completion, up to 24 months post-infusion
Total Hgb without disease-indicated transfusion support | through study completion, up to 24 months post-infusion
Change in annualized packed red blood cell (pRBC) transfusion requirements (volume and frequency) for SCD indications | through study completion, up to 24 months post-infusion
Proportion of participants with complete resolution of severe vaso-occlusive crises (sVOCs) | over time, from 6 months to 18 months post-infusion
Incidence rate of any sVOCs | over time, from 6 months to study completion, up to 24 months post-infusion
Proportion of participants achieving HbS <50% for at least 3 months | through study completion, up to 24 months post-infusion
Evaluation of globin chain expression compared to baseline | through study completion, up to 24 months post-infusion

CONTACTS AND LOCATIONS:
Overall Officials: Mathew Porteus, MD, PhD, Study Director — Kamau Therapeutics
Locations (4):
- United States (4):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Lucile Packard Children's Hospital, Palo Alto, California
  - Washington University, St Louis, Missouri
  - Nationwide Children's Hospital, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: Undecided